CLINICAL TRIAL: NCT06729073
Title: A Phase 1, Multiple-dose, Single-center, Randomized, Open-label, 2-period, 2-treatment Crossover Systemic Bioavailability Study of Diclofenac Comparing AMZ001 (Diclofenac Sodium Gel) Applied Once Daily on Each Knee Diclofenac Diethylammonium Gel 1.16% Applied 4 Times Daily on Each Knee in Healthy Subjects
Brief Title: Comparison of Diclofenac Systemic Exposure From Two Different Products (AMZ001 and Diclofenac Diethylammonium 1.16% Gel) in Healthy Participants After Repeated Topical Administrations for 7 Days.
Acronym: AMZ001
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amzell (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AMZ001-009
Record Dates: First submitted 2024-12-06; First posted 2024-12-11 (Actual); Results first posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Healthy Volunteer
Keywords: pharmacokinetics
MeSH Terms: interventions — diclofenac diethylamine; Gels

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AMZ001 (Experimental): AMZ001 applied once daily for 7 consecutive days
  Interventions: Drug: Diclofenac sodium gel
- Diclofenac diethylamine 1.16% (Active Comparator): Reference product applied four-times daily for 7 consecutive days
  Interventions: Drug: Diclofenac diethylamine 1.16% gel

INTERVENTIONS:
Drug: Diclofenac sodium gel — topical administration
  Arms: AMZ001
Drug: Diclofenac diethylamine 1.16% gel — Topical administration
  Arms: Diclofenac diethylamine 1.16%

SUMMARY:
The aim of the present study is to investigate the systemic bioavailability of AMZ001, applied once daily on each knee compared to Diclofenac diethylammonium gel 1.16%, applied 4 times daily on each knee, after repeated dosing in healthy subjects for 7 days The safety and local tolerability of AMZ001, applied once daily, will be evaluated after repeated dosing in healthy subjects for 7 days

DETAILED DESCRIPTION:
On their both knees, participants will apply once daily AMZ001 for 7 consecutive days. Participants will also apply Diclofenac Diethylammonium 1.16% Gel as per label information on each knee.

Intensive pharmacokinetic assessment (blood samplings) will be performed on the first day of application (Day 1) as well as on the last day of application (Day 7).

Each participant will receive each of the two treatments in a randomized manner. Between each treatment, participant will not receive any of tested therapies during at least 21 days before receiving the next therapy. (washout period)

Participants will stay on the clinical unit only during each period of treatment but not during washout period.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) within the range of 18.0-30.0 kg/m^2 (inclusive) at screening
* Female participant is eligible to participate if she is not pregnant or breastfeeding, and one of the following conditions applies:

  * Is a WONCBP. A WOCBP must have a negative highly sensitive serum pregnancy test at screening OR
  * Is a WOCBP and using a contraceptive method that is highly effective (with a failure rate of <1% per year), preferably with low user dependency, without interruption, during trial participation and until 30 days after the last administration of study intervention and agrees not to donate eggs (ova, oocytes) for the purpose of reproduction during this period.
* Participant is overtly healthy as determined by medical evaluation including medical history, full physical examination, vital signs, and ECG
* Participant is free of any systemic or dermatologic disorder and chronic or acute infections, which, in the opinion of the Investigator, may interfere with the study results or increase the risk of adverse events.
* Participant is a non-smoker, former smoker or stable non-smoker (= 0 cigarettes, pipes, cigars, or others) for at least 3 months prior to screening. Participant must also have abstained from use of other nicotine containing products (e.g., nicotine patch, chewing gum or e-cigarettes) for at least 3 months before screening.
* Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the ICF and in this protocol prior to any clinical study specific procedure.

Exclusion Criteria:

* Any visible skin disease, skin lesions, wounds, or a significant amount of hair at the application sites (both knees).
* Any history or evidence of any clinically relevant cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrinologic, hematologic, immunologic, metabolic, genitourinary, pulmonary, neurologic, dermatologic, musculoskeletal, psychiatric and/or other major disease as determined by medical evaluation (including [abbreviated] physical examination) capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study intervention; or interfering with the interpretation of data.
* Any known or suspected malignancy, excluding basal cell cancer unless it is associated with the treatment area.
* Any gastrointestinal bleeding issues, e.g., Gastroesophageal Reflux Disease, Peptic Ulcer Disease.
* Any hospital admission or major surgery within 30 days prior to randomization
* History or current evidence of ongoing hepatic disease or impaired hepatic function at screening as indicated by diagnostic assessments
* History or current evidence of renal disease or impaired renal function at screening as indicated by diagnostic assessments
* Any clinically relevant history of allergic conditions requiring hospitalization or prolonged systemic treatment (including drug allergies, drug hypersensitivity, asthma, angioedema, urticaria, eczema, acute rhinitis precipitated by acetylsalicylic acid or other NSAIDs, allergies requiring therapy with corticosteroids or anaphylactic reactions), excluding allergic contact sensitizations (e.g., nickel allergy). Subjects with uncomplicated seasonal allergic rhinitis can be accepted only if the expected allergy season is clearly outside enrolment/ treatment periods.
* Known or suspected hypersensitivity to diclofenac, or any components of the formulations used
* Contraindications for the use of study interventions
* Any clinically relevant chronic or acute infectious illnesses or febrile infections within 2 weeks prior to the first scheduled administration of study intervention
* Evidence of COVID-19 signs or symptoms or confirmed COVID-19 infection within the last 2 weeks prior to screening.
* Treatment with systemic or local diclofenac within 30 days of enrollment or during the study (except for study interventions).
* Use of any concomitant medication or any drugs / medicines (including over-the-counter medication, dietary supplements, natural and herbal remedies) within 2 weeks before the first scheduled administration of study intervention or within less than 10 times the elimination half-life of the respective drug (whichever is longer) or is anticipated to require concomitant medication during the 2-week period or at any time throughout the study.
* Use of any topical medication, cosmetics, cream, ointments, lotions on the treatment site 2 weeks prior to enrollment through EOT visit.
* Use of any investigational drug or participation in any clinical study within 30 days or 10 half-life times (if known) of study drug administered in a previous trial, whichever is longer, prior to the expected date of first administration of study intervention.
* Positive for hepatitis B surface antigen (HBsAg), hepatitis C virus antibodies (anti-HCV) and anti-human immunodeficiency virus antibodies (anti-HIV 1 and 2 and HIV 1-p24 antigen) at screening
* Positive screen for alcohol, drugs of abuse and cotinine test at screening.
* Female subject who plans to become pregnant during the clinical study period and for 3 months after final study intervention administration
* Donation or blood collection of more than 1 unit (approximately 450 mL) of blood (or blood products) or acute loss of blood during the 30 days prior to randomization.
* Employee of the Sponsor, or Contract Research Organization (CRO) involved in the clinical study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2024-11-29 (Actual); Primary Completion 2025-06-10 (Actual); Study Completion 2025-07-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Nuvisan, Neu-Ulm, Germany

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- AMZ001/Diclofenac Diethylamine 1.16%: AMZ001 applied once daily for 7 consecutive days followed by at least 21-day washout followed by Diclofenac diethylamine 1.16% applied four times daily for 7 consecutive days
- Diclofenac Diethylamine 1.16%/AMZ001: Reference product applied four-times daily for 7 consecutive days followed by at least 21-day washout followed by AMZ001 applied once daily for 7 consecutive days
Period: 1
Arm/Group | AMZ001/Diclofenac Diethylamine 1.16% | Diclofenac Diethylamine 1.16%/AMZ001
Started | 17 | 17
Completed | 17 | 17
Not Completed | 0 | 0
Period: 2
Arm/Group | AMZ001/Diclofenac Diethylamine 1.16% | Diclofenac Diethylamine 1.16%/AMZ001
Started | 17 | 16
Completed | 17 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AMZ001/Diclofenac Diethylamine 1.16% | Diclofenac Diethylamine 1.16%/AMZ001 | Total
Number analyzed (Participants) | 17 | 17 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.2 (12.75) | 44.5 (9.94) | 45.8 (11.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 7 | 18
  Male | 6 | 10 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 17 | 15 | 32
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 17 | 34
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve 0-24h
Description: Area under the curve from time zero to 24 hours
Time Frame: Day 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | AMZ001 | Diclofenac Diethylamine 1.16%
Number analyzed (Participants) | 33 | 34
h*ng/mL | 281.60 (67.1) | 411.35 (57.2)

2. Secondary Outcome: Pharmacokinetic Parameter - Cmin
Description: Minimum plasma drug concentration (Cmin)
Time Frame: Day 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | AMZ001 | Diclofenac Diethylamine 1.16%
Number analyzed (Participants) | 33 | 34
ng/mL | 5.812 (73.1) | 10.22 (50.2)

3. Secondary Outcome: Pharmacokinetic Parameter - Cavg
Description: Average plasma concentration (Cavg)
Time Frame: Day 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | AMZ001 | Diclofenac Diethylamine 1.16%
Number analyzed (Participants) | 33 | 34
ng/mL | 11.733 (67.1) | 17.139 (57.2)

4. Secondary Outcome: Pharmacokinetic Parameter - Tmax
Description: Time to reach maximum plasma concentration (Tmax)
Time Frame: Day 7
Measure: Median (Full Range); unit: h
Arm/Group | AMZ001 | Diclofenac Diethylamine 1.16%
Number analyzed (Participants) | 33 | 34
h | 6 [0 to 20.017] | 17.9830 [0 to 24]

5. Secondary Outcome: Compare Exposure to Diclofenac
Description: Area under the curve from time zero to 24 hours and maximum (peak) plasma drug concentration
Time Frame: Day 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | AMZ001 | Diclofenac Diethylamine 1.16%
Number analyzed (Participants) | 33 | 34
h*ng/mL | 141.76 (101.6) | 86.76 (116.3)

6. Secondary Outcome: Pharmacokinetic Parameter - Tmax
Description: Time to reach maximum plasma concentration (Tmax)
Time Frame: Day 1
Measure: Median (Full Range); unit: h
Arm/Group | AMZ001 | Diclofenac Diethylamine 1.16%
Number analyzed (Participants) | 33 | 34
h | 9.9170 [4.000 to 23.833] | 23.8330 [8.000 to 23.883]

7. Secondary Outcome: Pharmacokinetic Parameter - Cavg
Description: Average plasma concentration
Time Frame: Day 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | AMZ001 | Diclofenac Diethylamine 1.16%
Number analyzed (Participants) | 33 | 34
ng/mL | 5.906 (101.6) | 3.615 (116.3)

8. Secondary Outcome: Incidence of Application Site Reactions
Description: Number of subjects having at least one event
Time Frame: Day 1 to Day 7
Measure: Count of Participants; unit: Participants
Arm/Group | AMZ001 | Diclofenac Diethylamine 1.16%
Number analyzed (Participants) | 33 | 34
Participants | 0 | 1

ADVERSE EVENTS:
Time Frame: From enrollment until end of treatment period 2
Arm/Group | AMZ001 | Diclofenac Diethylamine 1.16%
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/34
Other Adverse Events (participants affected / at risk) | 5/33 | 8/34
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AMZ001 (N=33) | Diclofenac Diethylamine 1.16% (N=34)
Nasopharyngitis (Infections and infestations) | 2 | 3
Rhinitis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Headache (Nervous system disorders) | 1 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol (2024-10-10): https://cdn.clinicaltrials.gov/large-docs/73/NCT06729073/Prot_000.pdf